CLINICAL TRIAL: NCT02413203
Title: A Randomized, Double-blinded, Placebo-controlled Study Investigating the Pharmacological Response to Celecoxib Using ex Vivo Human Whole-blood Assay (hWBA) and Broad-spectrum Lipidomics Analysis
Brief Title: Lipidomics Screening of Celecoxib in ex Vivo Human Whole Blood Assay - Part B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: 818658-Part B
Record Dates: First submitted 2015-03-19; First posted 2015-04-09 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Healthy
Keywords: lipidomics; ex vivo human whole blood assay; celecoxib; selective COX-2 inhibitor
MeSH Terms: interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Celecoxib (Experimental): Oral administration of a single pill of celecoxib (200 mg). Celecoxib pills will be over-encapsulated to match the placebo.
  Interventions: Drug: Celecoxib
- Placebo (Placebo Comparator): Oral administration of a single placebo pill.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib — Blood and urine collections before and 3 hours after celecoxib administration.
  Other Names: Celebrex
  Arms: Celecoxib
Drug: Placebo — Blood and urine collections before and 3 hours after placebo administration.
  Arms: Placebo

SUMMARY:
Cardiovascular complications of NSAIDs, selective for inhibition of COX-2, stimulated interest in microsomal prostaglandin E synthase-1 (mPGES-1) as an alternative drug target. Global deletion of mPGES-1 in mice suppresses prostaglandin (PG) E2 and augments PGI2 by PGH2 substrate rediversion. Unlike COX-2 inhibition or gene deletion, mPGES-1 deletion does not cause a predisposition to thrombogenesis and hypertension. However, cell-specific deletion of mPGES-1 reveals that the predominant substrate rediversion product among the prostaglandins varies by cell type, complicating drug development. The research team has developed an ultra performance liquid chromatography/ tandem mass spectrometry (UPLC-MS/MS) technique that allows the quantification of a wide range of lipids beyond the prostaglandin pathway (leukotrienes, anandamide and the 2-arachidonylglycerol cascades).

This study is designed to examine different pathway interventions from the arachidonic acid cascade by anti-inflammatory compounds (with a focus on mPGES-1 inhibition) in whole human blood in vitro (Part A) and ex vivo (Part B). In Part B, healthy volunteers will be asked to take a single, therapeutic dose of celecoxib and blood and urine samples will be collected before and after drug administration. Collected blood will be stimulated ex vivo, and lipids and their metabolites will be measured in blood and urine, respectively. The investigators expect that lipid profile from ex vivo hWBA done on celecoxib-treated subjects will recapitulate findings from the in vitro hWBA received with celecoxib-treated human blood (Part A).

DETAILED DESCRIPTION:
Nonsteroidal anti-inflammatory drugs (NSAIDs), selective for inhibition of cyclooxygenase (COX)-2, alleviate pain and inflammation by suppressing COX-2-derived prostacyclin (PGI2) and prostaglandin (PG) E2 (1). However, eight placebo-controlled clinical trials have revealed that NSAIDs, designed to inhibit specifically COX-2, predispose patients to increased cardiovascular risks including myocardial infarction, stroke, systemic and pulmonary hypertension, congestive heart failure, and sudden cardiac death (1-3). The cardiovascular adverse effects are attributable to the suppression of COX-2-derived PGI2, a potent vasodilator and inhibitor of platelet activation (4; 5). The research team has shown that global deletion, selective inhibition or mutation of COX-2, or deletion of the receptor for PGI2 elevate blood pressure and accelerate thrombogenesis in mouse models (6). The investigators have further demonstrated that vascular COX-2 deletion predisposes mice to thrombosis and hypertension (7), and that selective deletion of COX-2 in cardiomyocytes leads to cardiac dysfunction and enhanced susceptibility to induced arrhythmogenesis (8) that may contribute to the heart failure and cardiac arrhythmias reported in patients taking NSAIDs specific for inhibition of COX-2.

This cardiovascular hazard from NSAIDs prompted interest in the microsomal prostaglandin E synthase-1 (mPGES-1) as an alternative drug target. mPGES-1 is the inducible PG terminal synthase that acts downstream of COX-2 and catalyzes the conversion of the intermediate COX endoperoxide product PGH2 to PGE2 (9). The investigators have previously reported that similar to the interference with COX-2 expression or function, global or cell-specific deletion of mPGES-1 suppresses PGE2 production; but unlike with COX-2, global mPGES-1 deficiency augments biosynthesis of PGI2 and does not predispose normo- or hyperlipidemic mice to thrombogenic or hypertensive events (9-11). Both suppression of PGE2 and augmentation of PGI2 in mPGES-1-/- mice result from the rediversion of the accumulated PGH2 substrate to PGI2 synthase (10). Furthermore, global deletion of mPGES-1 limits the vascular proliferative response to wire injury (12), retards atherogenesis and suppresses angiotensin II-induced abdominal aortic aneurysm formation in hyperlipidemic mice (10; 13). The research team has also shown that mPGES-1-deficiency does not affect ozone-induced airway inflammation or airway hyper-responsiveness suggesting that pharmacological inhibition of mPGES-1 and endoperoxide rediversion to PGD2 may not predispose patients at risk to airway dysfunction (14). In addition, studies by others indicate that global deletion of mPGES-1 reduces the post-ischemic brain infarction and neurological dysfunction in cerebral ischemia/reperfusion in mice (15). mPGES-1 deficiency also renders mice less susceptible to excessive inflammation and hypersensitivity in rodent models of analgesia (16; 17). Taken together, these findings suggest that pharmacological inhibition of mPGES-1 may retain anti-inflammatory effects from PGE2 suppression, but due to PGI2 augmentation, targeting of mPGES-1 might avoid the cardiovascular risks associated with selective COX-2 inhibitors.

PGH2 substrate rediversion consequent to mPGES-1 deletion is a ubiquitous event observed at the cellular level and systemically (urinary prostaglandin metabolites); the profile of the rediversion products, however, varies by cell and tissue type, the disease model, and the extent of system perturbation (6; 10-14; 18-21). The investigators have shown that in mice deficient in mPGES-1 in endothelial cells (EC) or vascular smooth muscle cells (VSMC), PGI2 is the predominant substrate rediversion product, whereas deletion of mPGES-1 in myeloid cells results in shunting of PGH2 mostly towards TxA2(11). Functionally, mice lacking mPGES-1 in myeloid cells, exhibited a poor response to vascular injury implicating myeloid mPGES-1 as a cardiovascular drug target. Therefore, cell-specific mPGES-1 deletion leads to a differential pattern of substrate rediversion and may affect biological function of the system, thus complicating drug development. What is unknown is whether genetic deletion or pharmacological inhibition of mPGES-1 can directly (through substrate rediversion) or indirectly (by effects of prostaglandin rediversion products on enzyme expression or their further metabolism to transcellular products (22)) influence the lipidome beyond the prostaglandin pathway with functional consequence. For example, disruption of AA-PGE2 metabolism might influence arachidonate product formation by the cytochrome P450 (23; 24), leukotriene, anandamide, 2-arachidonylglycerol (2-AG) and other cascades (25). At the cellular level, mPGES-1-/- macrophages, pretreated with LPS and stimulated with arachidonic acid (AA), exhibit a 5-fold increase in 12-HHT (12-hydroxyheptadecatrienoic acid), indicating substrate rediversion towards thromboxane A synthase (18). Inhibition and deletion of COX-2 have been reported to augment metabolites of 5-lipoxygenase (5-LO) pathway 5-HETE (5-hydroxyeicosatetraenoic acid) and leukotrienes LTB4, LTC4, LTD4 (26-28), and metabolites of CYP450 cascade 14,15-DHET/EET (dihydroxyeicosatrienoic/epoxyeicosatrienoic acid) (26). Therefore, the substrate AA may be shunted from one pathway to the other when a particular branch of the cascade is pharmacologically inhibited or genetically ablated.

Here, the research team will conduct a broad-spectrum lipidomics screening of anti-inflammatory drugs and drug candidates that antagonize receptors (LTC4, LTB4, EP4 receptors) or inhibit specific components (COX-1, COX-2, mPGES-1, 5-KO, FLAP, LTA4A) of arachidonic acid pathway in an in vitro human whole-blood assay (hWBA).

Preliminary in vitro results from Part A demonstrated that targeting of COX-2 with a selective COX-2 inhibitor celecoxib affected not only cyclooxygenase pathway but also lipoxygenase cascade. Celecoxib inhibited COX-derived products PGE2, PGF2a and TxB2 and significantly reduced levels of 15-HETE, a product of 15-LOX cascade.

In Part B, the investigators propose to study the effect of celecoxib on plasma lipids ex vivo. Healthy, non-smoking, male and female volunteers will be asked to take a single, therapeutic dose of 200 mg of celecoxib or a placebo pill and provide blood and urine samples before and after the drug administration. Experiments will include (i) the ex vivo whole blood assay, in which lipids will be measured in blood collected before and 3 hours (Tmax) after administration of celecoxib and stimulated with LPS, (ii) lipid metabolites will be measured in pre- and post-celecoxib urine samples, (iii) celecoxib plasma and urine concentrations will be measured to evaluate the pharmacokinetic profile of the study drug.

The investigators expect that lipid profile from ex vivo hWBA done on celecoxib-treated subjects will recapitulate findings from the in vitro hWBA received with celecoxib-treated human blood.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 - 50
* Volunteers must be in good health as based on medical history
* All volunteers must be non-smoking and non-pregnant

Exclusion Criteria:

* Subjects with any medical condition, which according to the investigator, may interfere with interpretation of the study results, be indicative of an underlying disease state, or compromise the safety of a potential subject (cancer or history of significant cardiovascular disease (including stroke or TIA), renal, hepatic, gastrointestinal, respiratory, endocrine, metabolic, hematopoietic, or neurological disorders).
* Subjects who have received an experimental drug within 30 days prior to the study
* Subjects who have taken medications at least two weeks prior to the study. Subjects using hormonal birth control, however, will not be an exclusionary criterion.
* Subjects who have taken aspirin or aspirin containing products for at least two weeks prior to the study.
* Subjects who are sensitive or allergic to celecoxib (Celebrex) or its components
* Subjects who have taken any formulation of celecoxib including but not limited to Celebrex, Celebra, Onsenal for at least two weeks prior to the start of the study and throughout the study
* Subjects who have taken acetaminophen, NSAIDs, COX-2 inhibitors (OTC or prescription) for at least two weeks prior to the study.
* Subjects who are consuming any type of tobacco product(s).
* Subjects who consume high doses of antioxidant vitamins daily (vitamin C> 1000mg, Vitamin E> 400IU, Beta Carotene> 1000IU, Vitamin A> 5000IU, Selenium> 200mcg, Folic Acid> 1mg) for the two weeks prior to the start of the study and throughout the study.
* Subjects who consume alcohol, caffeine or high fat food 24 hours prior to the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Garret FitzGerald, MD, Principal Investigator — University of Pennsylvania, Institute for Translationals Medicine and Therapeutics
Locations (1):
- The Clinical Translational Research Center (CTRC) at the Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Celecoxib | Placebo
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Celecoxib | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (8.6) | 30 (9) | 32.1 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Quantification of Plasma Lipids in the Whole Blood: Prostaglandin E2 (PGE2)
Description: PGE2 in blood taken from celecoxib-treated subjects and stimulated ex vivo with LPS was compared to similarly treated blood from placebo group. Plasma PGE2 was normalized to sample volume (ng/ml) and expressed as a percentage of subject's pre-dose control using the formula: percentage of pre-dose control = (Cpost-dose/Cpre-dose) × 100%, where C represents PGE2 concentration in ng/ml.
Time Frame: A single visit of around 4 hours
Measure: Mean (Standard Deviation); unit: percentage of pre-dose control
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 10 | 10
percentage of pre-dose control | 49.9 (26.59) | 110 (49.2)

2. Primary Outcome: Quantification of Plasma Lipids in the Whole Blood: Prostaglandin F2a (PGF2a)
Description: PGF2a in blood taken from celecoxib-treated subjects and stimulated ex vivo with LPS was compared to similarly treated blood from placebo group. Plasma PGF2a was normalized to sample volume (ng/ml) and expressed as a percentage of subject's pre-dose control using the formula: percentage of pre-dose control = (Cpost-dose/Cpre-dose) × 100%, where C represents PGF2a concentration in ng/ml.
Time Frame: A single visit of around 4 hours
Measure: Mean (Standard Deviation); unit: percentage of pre-dose control
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 10 | 10
percentage of pre-dose control | 45.48 (20.51) | 97.2 (32.9)

3. Primary Outcome: Quantification of Plasma Lipids in the Whole Blood: Thromboxane B2 (TxB2)
Description: TxB2 in blood taken from celecoxib-treated subjects and stimulated ex vivo with LPS was compared to similarly treated blood from placebo group. Plasma TxB2 was normalized to sample volume (ng/ml) and expressed as a percentage of subject's pre-dose control using the formula: percentage of pre-dose control = (Cpost-dose/Cpre-dose) × 100%, where C represents TxB2 concentration in ng/ml.
Time Frame: A single visit of around 4 hours
Measure: Mean (Standard Deviation); unit: percentage of pre-dose control
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 10 | 10
percentage of pre-dose control | 52.2 (16.9) | 83.4 (12.8)

4. Primary Outcome: Quantification of Plasma Lipids in the Whole Blood: 15-Hydroxyeicosatetraenoic Acid (15-HETE)
Description: 15-HETE in blood taken from celecoxib-treated subjects and stimulated ex vivo with LPS was compared to similarly treated blood from placebo group. Plasma 15-HETE was normalized to sample volume (ng/ml) and expressed as a percentage of subject's pre-dose control using the formula: percentage of pre-dose control = (Cpost-dose/Cpre-dose) × 100%, where C represents 15-HETE concentration in ng/ml.
Time Frame: A single visit of around 4 hours
Measure: Mean (Standard Deviation); unit: percentage of pre-dose control
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 10 | 10
percentage of pre-dose control | 49 (18.7) | 81.65 (22.8)

5. Secondary Outcome: Urinary Lipid Metabolites: PGE2 Metabolite (PGE-M)
Description: Effect of celecoxib on systemic PGE2 was assessed by comparing urine PGE-M in celecoxib vs placebo-treated groups. Urine data are reported as a percentage of the volunteer's own pre-dose control using the formula: percentage of pre-dose control = (Cpost-dose/Cpre-dose) × 100%, where C represents metabolite concentration in ng/mg creatinine.
Time Frame: A single visit of around 4 hours
Measure: Mean (Standard Deviation); unit: percentage of pre-dose control
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 10 | 10
percentage of pre-dose control | 79.15 (24.19) | 106 (20.1)

6. Secondary Outcome: Celecoxib Plasma Concentration
Description: Celecoxib plasma concentration will be measured in drug-treated and placebo groups by UPLC-MS/MS, and will be expressed as amount of the drug per volume of plasma (ng/ml). At Tmax of 3 hours after a single oral dose of celecoxib of 200 mg, drug plasma concentration should correspond to the maximum plasma concentration or Cmax.
Time Frame: A single visit of around 4 hours
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 10 | 10
ng/ml | 352.6 (221) | 0 (0)

7. Secondary Outcome: Urinary Lipid Metabolites: PGI2 Metabolite (PGI-M)
Description: Effect of celecoxib on systemic PGI2 was assessed by comparing urine PGI-M in celecoxib vs placebo-treated groups. Urine data are reported as a percentage of the volunteer's own pre-dose control using the formula: percentage of pre-dose control = (Cpost-dose/Cpre-dose) × 100%, where C represents metabolite concentration in ng/mg creatinine.
Time Frame: A single visit of around 4 hours
Measure: Mean (Standard Deviation); unit: percentage of pre-dose control
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 10 | 10
percentage of pre-dose control | 41.47 (11) | 78.6 (52.23)

8. Secondary Outcome: Urinary Lipid Metabolites: TxB2 Metabolite (Tx-M)
Description: Effect of celecoxib on systemic TxB2 was assessed by comparing urine Tx-M in celecoxib vs placebo-treated groups. Urine data are reported as a percentage of the volunteer's own pre-dose control using the formula: percentage of pre-dose control = (Cpost-dose/Cpre-dose) × 100%, where C represents metabolite concentration in ng/mg creatinine.
Time Frame: A single visit of around 4 hours
Measure: Mean (Standard Deviation); unit: percentage of pre-dose control
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 10 | 10
percentage of pre-dose control | 79 (14.4) | 77.9 (17.2)

ADVERSE EVENTS:
Arm/Group | Celecoxib | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No